CLINICAL TRIAL: NCT02281344
Title: A Proof-of-concept Study to Assess the Effect of MMV390048 Against Early Plasmodium Falciparum Blood Stage Infection in Healthy Participants.
Brief Title: MMV390048 Against Early Plasmodium Falciparum Blood Stage Infection in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inconsistent and unpredictable exposures were observed. Drug needed to be reformulated.
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Q-Pharm Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: QP14C11
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Malaria, Falciparum
Keywords: induced blood stage malaria infection
MeSH Terms: conditions — Malaria, Falciparum | interventions — MMV390048

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cohort 1 (Experimental): Cohort 1 will receive a single dose of 20mg MMV390048.
  Interventions: Drug: MMV390048 20mg

INTERVENTIONS:
Drug: MMV390048 20mg — Supplied as a powder to be prepared as a suspension for oral use

SUMMARY:
A single-centre, open-label, study using induced blood stage malaria infection to characterize the activity of MMV390048 against early Plasmodium falciparum blood stage infection.

DETAILED DESCRIPTION:
Study using induced blood stage malaria infection to characterize the activity of MMV390048 against early Plasmodium falciparum blood stage infection. There will be two or more cohorts of 8 subjects. In the first cohort a single dose of 20 mg of MMV390048 will be investigated. Depending on the data obtained, the dose in Cohort 2 may be adjusted but will not exceed the maximum tolerated dose (or highest achieved dose based on a predefined exposure cap) as determined in an ongoing single ascending dose study. Each participant will be inoculated on Day 0 with ~1,800 viable parasites of Plasmodium falciparum-infected human erythrocytes intravenously. On an outpatient basis, participants will be monitored daily until positive for presence of malaria parasites. Once positive they will be monitored twice-daily until treatment, for adverse events and the unexpected early onset of symptoms, signs or parasitological evidence of malaria. On the day designated for commencement of treatment, participants will be admitted to the study unit and monitored. The threshold for commencement of treatment will be when quantification of all participants is ≥ 1,000 parasites/mL. If the quantification of any participant is ≥ 5,000 parasites/mL, and is accompanied by a clinical symptom score >5, or if clinical or parasitological evidence of malaria occurs in any participant before all participants have reached the treatment threshold (quantification of ≥ 1,000), then treatment of that participant will begin within a 24 h period.

Following treatment with MMV390048, participants will be followed up as inpatients for at least 72 hours to ensure tolerance of the treatment and clinical response, then on an outpatient basis if clinically well for monitoring of safety and clearance of malaria parasites. Compulsory treatment with Riamet® (artemether-lumefantrine) will start on day 16 (±3 days) post study treatment unless required earlier. Early intervention can occur if either poor responses or fast responses are seen following MMV390048 treatment. This is to ensure participant safety and to avoid participant inconvenience if useful data cannot be obtained. Pre-emptive treatment with Riamet® can commence whenever necessary. Participants will be treated with a single dose (45 mg) of primaquine (Primacin™) at the end of their Riamet® treatment if gametocytes are identified, to ensure complete clearance of any gametocytes present.

ELIGIBILITY:
Inclusion Criteria:

* Participants who do not live alone from Day 0 until at least the end of the antimalarial drug treatment, and are contactable and available for the duration of the trial (≤4 months)
* Body weight ≥50kg, body mass index between 18.0 and 32.0 kg/m2, inclusive
* Healthy by clinical assessment
* Normal vital signs
* Normal 12-lead electrocardiogram
* Lab tests in normal range
* Agrees to use a double barrier method of contraception including condom plus diaphragm or condom plus intrauterine device or condom plus stable oral / transdermal / injectable hormonal contraceptive by female partner for ≥14 days prior to the first dose of study drug until 90 days after the last dose
* Written informed consent before any study procedure

Exclusion Criteria:

* History of malaria or participation in a previous malaria challenge study
* Must not have travelled to or lived >2 weeks in a malaria-endemic area in past 12 months nor plan to travel to one during study
* Evidence of increased cardiovascular disease risk
* History of splenectomy
* Presence / history of drug hypersensitivity, or allergic disease diagnosed and treated or history of a severe allergic reaction, anaphylaxis or convulsions following any vaccination or infusion
* Presence of current / suspected serious chronic diseases such as cardiac or autoimmune disease, diabetes, progressive neurological disease, severe malnutrition, acute or progressive hepatic or renal disease, psoriasis, rheumatoid arthritis, asthma, epilepsy or obsessive compulsive disorder, skin carcinoma excluding non-spreadable skin cancers such as basal cell and squamous cell carcinoma, schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis
* History of photosensitivity
* History of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis, including depression or receiving psychiatric drugs or hospitalized in past 5 yrs for psychiatric illness, history of suicide attempt or confinement for danger to self/others
* Frequent headache and/or migraine, recurrent nausea, and/or vomiting (≥2 / month)
* Acute infectious disease/fever in 5 days pre-inoculation with malaria parasites
* Acute illness in 4 weeks pre-screening which may compromise subject safety
* Any significant intercurrent disease, in particular liver, renal, cardiac, pulmonary, neurologic, rheumatologic, or autoimmune disease by history, physical exam or lab test
* Clinically significant disease or any condition that might affect drug absorption distribution or excretion
* Participation in any investigational study in last 12 weeks
* Any blood sampling/donation in last 8 weeks
* Unwilling to defer blood donation for 6 months
* Any blood donation, in 1 month before inclusion.
* Medical requirement for intravenous immunoglobulin or blood transfusion
* Ever had a blood transfusion
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension
* History or presence of alcohol abuse (≥40g per day) or drug habituation, or any prior intravenous use of an illicit substance
* Smoking ≥5 cigarettes or equivalent /day and unable to stop smoking during confinement period
* Poppy seeds in 24h pre-screening
* Excessive consumption of xanthine bases, including red bull, chocolate
* Any medication (including St John's Wort) in 14 days pre-study or within 5 times the medication half-life if longer
* Vaccination in the last 28 days
* Any corticosteroids, anti-inflammatory, immunomodulators or anticoagulants. Any currently or previous immunosuppressive therapy, including systemic steroids including adrenocorticotrophic hormone or inhaled steroids in dosages associated with hypothalamic-pituitary-adrenal axis suppression or chronic use of inhaled high potency corticosteroids
* Recent or current systemic therapy with an antibiotic / potential antimalarial
* Likely to be noncompliant, or unable to cooperate
* Not contactable in case of emergency throughout and for 2 weeks after end of study
* Staff directly involved in study conduct
* Without good peripheral venous access
* Positive for: hepatitis B surface antigen, anti-hepatitis B core antibodies, anti-hepatitis C virus antibodies, or anti-human immunodeficiency virus 1/2 antibodies
* glucose-6-phosphate dehydrogenase deficiency
* Positive urine drug screen or alcohol urine or breath test
* Cardiac/QT risk: Known pre-existing prolongation of the QTcB/QTcF interval considered clinically significant. Family history of sudden death or of congenital prolongation of the corrected QT interval interval or known congenital prolongation of the corrected QT interval or any clinical condition known to prolong the corrected QT interval interval. History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia. Electrolyte disturbances, particularly hypokalaemia, hypocalcaemia or hypomagnesaemia. Clinically relevant 12-lead electrocardiogram abnormality at screening or which will interfere with the analysis, or history of clinically significant abnormalities
* Known hypersensitivity to MMV390048 or any of its excipients or 4-aminoquinolines, artemether or other artemisinin derivatives, lumefantrine, or other arylaminoalcohols
* Unwillingness to abstain from citrus (grapefruit, Seville orange, etc.) or juice, as well as quinine containing foods/beverages for the study period
* Lactose intolerance
* Unwilling to restrict exposure to direct sunlight during the study. Must use sunglasses and sunblock for the study period

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2014-12-19 (Actual); Study Completion 2014-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McCarthy, Dr., Principal Investigator — Q-Pharm Pty Limited
Locations (1):
- Q-Pharm Clinics, Royal Brisbane and Women's Hospital, Brisbane, Queensland, Australia

REFERENCES:
- [Derived] Sinxadi P, Donini C, Johnstone H, Langdon G, Wiesner L, Allen E, Duparc S, Chalon S, McCarthy JS, Lorch U, Chibale K, Mohrle J, Barnes KI. Safety, Tolerability, Pharmacokinetics, and Antimalarial Activity of the Novel Plasmodium Phosphatidylinositol 4-Kinase Inhibitor MMV390048 in Healthy Volunteers. Antimicrob Agents Chemother. 2020 Mar 24;64(4):e01896-19. doi: 10.1128/AAC.01896-19. Print 2020 Mar 24. PMID 31932368
- [Derived] Burel JG, Apte SH, McCarthy JS, Doolan DL. Plasmodium vivax but Not Plasmodium falciparum Blood-Stage Infection in Humans Is Associated with the Expansion of a CD8+ T Cell Population with Cytotoxic Potential. PLoS Negl Trop Dis. 2016 Dec 8;10(12):e0005031. doi: 10.1371/journal.pntd.0005031. eCollection 2016 Dec. PMID 27930660

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 MMV390048 20mg: Cohort 1 will receive a single, dose of 20mg MMV390048.
  MMV390048 20mg: Supplied as a powder to be prepared as a suspension for oral use.
  The study was conducted in one cohort (n=6) using a 20 mg dose of MMV390048 Powder In Bottle (PIB). Dose escalation was planned in a subsequent cohort, but due to the inconsistent pharmacokinetic profiles of the PIB formulation it was decided to reformulate the compound before proceeding with the study.
Period: Overall Study
Arm/Group | Cohort 1 MMV390048 20mg
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1 MMV390048 20mg
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (4.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.50 (4.767)

OUTCOME MEASURES:

1. Primary Outcome: MMV390048 Area Under the Plasma Concentration Versus Time Curve (AUClast) up to Day 21 Post-dose
Description: Pharmacokinetic-pharmacodynamic relationship of MMV390048 on clearance of Plasmodium falciparum parasites from the blood in healthy participants following infection with blood stage parasites.
  The area under the plasma concentration time curve from time zero to the last measured time point.
Time Frame: At pre-dose, and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24 (D1), 30, 36, 48 (D2), 72 (D3), and 144 hours (D6) and Days 8, 10, 14, 18 and D21.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1 MMV390048 20mg
Number analyzed (Participants) | 6
ng*hr/mL | 9487 (2444)

2. Secondary Outcome: Parasite Reduction Rate (PRR) Following MMV390048 Treatment
Description: The clearance of malaria parasitemia by Polymerase Chain Reaction (PCR) measurement.
Time Frame: From dosing up to Day 21 Post-dose
Reporting Status: Not Posted

3. Secondary Outcome: MMV390048 Maximum Plasma Concentration (Cmax)
Description: Maximum Plasma Concentration (Cmax) of MMV390048
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 MMV390048 20mg
Number analyzed (Participants) | 6
ng/mL | 113 (43.8)

4. Secondary Outcome: MMV390048 Time to Maximum Plasma Concentration (Tmax)
Description: Time to Maximum Plasma Concentration (Tmax) of MMV390048
Time Frame: From dosing up to Day 21 Post-dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to Day 21 Post-dose
Arm/Group | Cohort 1 MMV390048 20mg
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 MMV390048 20mg (N=6)
Nausea (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (2)
Hot flush (General disorders) | 1 (1)
Hyperhidrosis (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (7)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (6)
Paraesthesia (Nervous system disorders) | 1 (1)
Rinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Dose escalation was planned for more than 1 cohort, but due to inconsistent pharmacokinetic profiles the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No